CLINICAL TRIAL: NCT00874016
Title: A Comparison of the Airtraq and Standard Direct Laryngoscopy in the Pediatric Airway - A Randomized Trial.
Brief Title: Airtraq Versus Standard Direct Laryngoscopy in the Pediatric Airway
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IWK Health Centre (Other)
Responsible Party: Arnim Vlatten, MD, Department of Pediatric Anesthesia, IWK Health Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Airtraq 4469
Record Dates: First submitted 2009-04-01; First posted 2009-04-02 (Estimated); Last update posted 2010-12-16 (Estimated); Status verified 2009-04

CONDITIONS: Endotracheal Intubation
Keywords: intubation; Airtraq; pediatric; airway

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Airtraq (Active Comparator): Intubation with the use of the Airtraq
  Interventions: Device: Airtraq
- Direct Laryngoscopy (Active Comparator): Intubation using direct laryngoscopy
  Interventions: Device: Direct Laryngoscopy

INTERVENTIONS:
Device: Airtraq — Intubation using Airtraq
  Arms: Airtraq
Device: Direct Laryngoscopy — Intubation using direct laryngoscopy
  Arms: Direct Laryngoscopy

SUMMARY:
Time to intubate, view to glottic opening and success rate are not different when Airtraq technique is used compared to standard direct laryngoscopy in children.

DETAILED DESCRIPTION:
50 children (age 5 years and 11 month or younger) with expected easy intubation, scheduled for elective surgery requiring endotracheal intubation are enrolled.

ELIGIBILITY:
Inclusion Criteria:

* elective surgery requiring endotracheal intubation

Exclusion Criteria:

* predicted difficult bag-mask ventilation
* predicted difficult intubation
* rapid sequence induction
* emergency endotracheal intubation
* hemodynamic instability
* emergency surgery
* non-english speaking caregivers/parents

Max Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2009-04; Primary Completion 2009-08 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Time to intubation | 1 day

SECONDARY OUTCOMES:
Percentage of glottic opening seen | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Arnim Vlatten, MD, Principal Investigator — IWK Health Centre
Locations (1):
- Department of Pediatric Anesthesia, IWK Health Centre, Halifax, Nova Scotia, Canada

REFERENCES:
- [Background] Maharaj CH, Costello JF, Harte BH, Laffey JG. Evaluation of the Airtraq and Macintosh laryngoscopes in patients at increased risk for difficult tracheal intubation. Anaesthesia. 2008 Feb;63(2):182-8. doi: 10.1111/j.1365-2044.2007.05316.x. PMID 18211450
- [Background] Maharaj CH, O'Croinin D, Curley G, Harte BH, Laffey JG. A comparison of tracheal intubation using the Airtraq or the Macintosh laryngoscope in routine airway management: A randomised, controlled clinical trial. Anaesthesia. 2006 Nov;61(11):1093-9. doi: 10.1111/j.1365-2044.2006.04819.x. PMID 17042849